CLINICAL TRIAL: NCT00256646
Title: CSP #465D - Markers And Mechanisms of Vascular Disease in Type II Diabetes
Brief Title: Markers and Mechanisms of Vascular Disease in Type II Diabetes
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 465D
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — samples without DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Patients who are enrolled in the ongoing randomized clinical trial AGlycemic Control and Complications in Diabetes Mellitus Type 2".
  Interventions: Drug: Rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone — ROSIGLITAZONE (roe si GLI ta zone) helps to treat type 2 diabetes. It helps to control blood sugar. Treatment is combined with diet and exercise.

SUMMARY:
OBJECTIVES: Vascular Disease is the leading cause of complications and death in patients with diabetes. Risk markers and underlying mechanisms have not been fully elucidated, and may differ from those in non-diabetic individuals. The unifying theme for the Program Project is that hyperglycemia and insulin resistance alter a number of biological processes which interact in vicious cycles to accelerate atherogenesis and are consequently major underlying risk factors for vascular disease. The overall objectives are to define these unique processes and to elucidate underlying biochemical, metabolic, and genetic determinants of vascular disease complications in diabetes.

RESEARCH PLAN: Over the past 4 years, we have collaborated with the DCCT/EDIC Study Group, and have made novel observations regarding vascular disease pathogenesis in Type 1 Diabetes. This work has focused our studies on specific pathogenic processes. We will now study a Type 2 Diabetes cohort from the VA Cooperative Study, "Glycemic Control and the Complications of Diabetes, Type 2", with high vascular disease event rates. These collaborations provide a unique opportunity to address the pathogenesis of accelerated atherogenesis in the two main types of diabetes, and will greatly augment the scientific knowledge that will be gained in the conduct of these world-class prospective trials.

METHODS: The Program Project has 4 projects and 3 cores. Project 1 will assess lipoproteins, glycoxidative stress, and inflammation as risk factors in studies involving Type 2 Diabetes patients and cultured cell systems. Based on preliminary data from our initial studies Type 1 patients, changes in the NMR lipoprotein subclass profile will be emphasized.

Project 2 will elucidate interactions between inflammation, modifications of lipoproteins, and autoimmunity in vascular disease risk. These novel concepts are also based upon exciting preliminary data pertaining to LDL-antibody complexes.

Project 3 will pursue interesting preliminary data and define the role of the kallikrein-kinin system in vascular disease complications, with effects on mitogenesis and matrix production.

Project 4 will assess the role of the Insulin Resistance Syndrome and novel factors secreted from adipocytes in the pathophysiology of biochemical risk factors and cardiovascular complications.

Cores include an Administrative Core, a Biostatistics and Epidemiology Core which will link with the trials data coordinating centers, and Molecular and Statistical Genetics Core. Investigators will work in close collaboration with the VA Executive Committee, Study Centers, the Hines Coordinating Center, and some of the other ancillary studies. All data analysis involving clinical outcomes will be performed at the Hines Coordinating Center.

There is true synergism among the projects at both scientific and logistical levels. The Program Project design allows for interactions among multidisciplinary investigators studying the same cohort, which will define how multiple pathological processes interact at the level of the arterial wall to promote atherosclerosis.

DETAILED DESCRIPTION:
Primary Hypothesis:

Secondary Hypotheses:

Primary Outcomes:

Study Abstract:

OBJECTIVES: Vascular Disease is the leading cause of complications and death in patients with diabetes. Risk markers and underlying mechanisms have not been fully elucidated, and may differ from those in non-diabetic individuals. The unifying theme for the Program Project is that hyperglycemia and insulin resistance alter a number of biological processes which interact in vicious cycles to accelerate atherogenesis and are consequently major underlying risk factors for vascular disease. The overall objectives are to define these unique processes and to elucidate underlying biochemical, metabolic, and genetic determinants of vascular disease complications in diabetes.

RESEARCH PLAN: Over the past 4 years, we have collaborated with the DCCT/EDIC Study Group, and have made novel observations regarding vascular disease pathogenesis in Type 1 Diabetes. This work has focused our studies on specific pathogenic processes. We will now study a Type 2 Diabetes cohort from the VA Cooperative Study, "Glycemic Control and the Complications of Diabetes, Type 2", with high vascular disease event rates. These collaborations provide a unique opportunity to address the pathogenesis of accelerated atherogenesis in the two main types of diabetes, and will greatly augment the scientific knowledge that will be gained in the conduct of these world-class prospective trials.

METHODS: The Program Project has 4 projects and 3 cores. Project 1 will assess lipoproteins, glycoxidative stress, and inflammation as risk factors in studies involving Type 2 Diabetes patients and cultured cell systems. Based on preliminary data from our initial studies Type 1 patients, changes in the NMR lipoprotein subclass profile will be emphasized.

Project 2 will elucidate interactions between inflammation, modifications of lipoproteins, and autoimmunity in vascular disease risk. These novel concepts are also based upon exciting preliminary data pertaining to LDL-antibody complexes.

Project 3 will pursue interesting preliminary data and define the role of the kallikrein-kinin system in vascular disease complications, with effects on mitogenesis and matrix production.

Project 4 will assess the role of the Insulin Resistance Syndrome and novel factors secreted from adipocytes in the pathophysiology of biochemical risk factors and cardiovascular complications.

Cores include an Administrative Core, a Biostatistics and Epidemiology Core which will link with the trials data coordinating centers, and Molecular and Statistical Genetics Core. Investigators will work in close collaboration with the VA Executive Committee, Study Centers, the Hines Coordinating Center, and some of the other ancillary studies. All data analysis involving clinical outcomes will be performed at the Hines Coordinating Center.

There is true synergism among the projects at both scientific and logistical levels. The Program Project design allows for interactions among multidisciplinary investigators studying the same cohort, which will define how multiple pathological processes interact at the level of the arterial wall to promote atherosclerosis.

Main Manuscript:

There is no independent data for this study, it was part of a larger study. Therefore there will be no results for this record/study.

ELIGIBILITY:
Inclusion Criteria:

Patients with type 2 DM who are no longer responsive to maximum dose of one or more oral agents

Exclusion Criteria:

Patients that did not participate in the VADT.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are enrolled in the ongoing randomized clinical trial AGlycemic Control and Complications in Diabetes Mellitus Type 2".
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is to define these unique processes and to elucidate underlying biochemical, metabolic, and genetic determinants of vascular disease complications in diabetes. | 2, 4, and 6 years.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Abraira, MD, Study Chair — Miami VA Healthcare System, Miami, FL
Locations (17):
- United States (16):
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, Tucson, Arizona
  - VA Central California Health Care System, Fresno, Fresno, California
  - VA Medical Center, Long Beach, Long Beach, California
  - VA San Diego Healthcare System, San Diego, San Diego, California
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - Richard Roudebush VA Medical Center, Indianapolis, Indianapolis, Indiana
  - VA Medical Center, Lexington, Lexington, Kentucky
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - VA Medical Center, Omaha, Omaha, Nebraska
  - VA New Jersey Health Care System, East Orange, East Orange, New Jersey
  - VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - VA South Texas Health Care System, San Antonio, San Antonio, Texas
  - VA Medical Center, Salem VA, Salem, Virginia
- VA Medical Center, San Juan, San Juan, Puerto Rico

REFERENCES:
- [Result] Lopes-Virella MF, Hunt KJ, Baker NL, Virella G, Moritz T; VADT Investigators. The levels of MDA-LDL in circulating immune complexes predict myocardial infarction in the VADT study. Atherosclerosis. 2012 Oct;224(2):526-31. doi: 10.1016/j.atherosclerosis.2012.08.006. Epub 2012 Aug 21. PMID 22963984
- [Result] Bhensdadia NM, Hunt KJ, Lopes-Virella MF, Michael Tucker J, Mataria MR, Alge JL, Neely BA, Janech MG, Arthur JM; Veterans Affairs Diabetes Trial (VADT) study group. Urine haptoglobin levels predict early renal functional decline in patients with type 2 diabetes. Kidney Int. 2013 Jun;83(6):1136-43. doi: 10.1038/ki.2013.57. Epub 2013 Mar 27. PMID 23536133